CLINICAL TRIAL: NCT05529901
Title: Post Marketing Surveillance of the GORE® CARDIOFORM Septal Occluder
Brief Title: Japan Post Marketing Surveillance of the GORE® CARDIOFORM Septal Occluder
Acronym: GSO-PFO PMS
Status: Active, not recruiting | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: JPS 21-08
Record Dates: First submitted 2022-08-23; First posted 2022-09-07 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Stroke; PFO - Patent Foramen Ovale; Cryptogenic Stroke; TIA
MeSH Terms: conditions — Stroke; Foramen Ovale, Patent; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: GORE® CARDIOFORM Septal Occluder — Patients for whom the device is used (implanted or used by not implanted) during the enrollment period of this post-marketing surveillance will be considered eligible for the study

SUMMARY:
The purpose of this post-marketing surveillance is to evaluate the effectiveness and safety of GORE® CARDIOFORM Septal Occluder under the post-marketing setting in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cryptogenic stroke (including transient ischemic attack with positive head imaging findings)
* Diagnosed with a PFO
* Note: Additional Inclusion Criteria may apply

Exclusion Criteria:

* N/A

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a cryptogenic stroke (including transient ischemic attack with positive head imaging findings) with possible involvement of patent foramen ovale (PFO) due to a presumed paradoxical embolism.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
PFO Closure Rate | 12 months
  PFO closure success will be defined as the number of cases which achieve effective PFO closure at 12 months post-initial procedure out of those which complete the PFO closure evaluation under Trans-Thoracic Echocardiography (TTE) with bubbles. PFO effective closure will be defined as the number of bubbles confirmed to be less than 20 (<20).
Rate of Conversion to surgical procedure | Discharge
  Rate of post-procedure conversion to surgical procedure will be calculated.
Incidence rate of post-procedure ischemic stroke events | 36 months
  Incidence rate of post-procedure ischemic stroke will be calculated. Additionally, those stroke events will be evaluated by Kapan-Meier plot.
Device success | 36 months
  Device success will be calculated by the number of cases with successful device implant during the initial procedure and later follow-ups out of those which underwent the transcatheter PFO closure procedure.
Incidence rate of post-procedure adverse events and/or device issues | 36 months
  Incidence rate of adverse events and/or device issues collected through each follow-up period will be calculated.
Incidence rate of device- and procedure-related events within 30 days post procedure | 30 days
  Incidence rate of adverse events and/or device issues which are defined as device- or procedure-related within 30 days post procedure will be calculated.

OTHER OUTCOMES:
Incidence rate of post-procedure Atrial fibrillation | 36 months
  Rate of post-procedure AF will be calculated during each follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Okayama University Hospital, Okayama, Japan

IPD SHARING:
Plan to Share IPD: No